CLINICAL TRIAL: NCT04898296
Title: Exploration of Possible Reasons for the Discrepancy Between Expectation and Indication of Subjective Perceived Exertions of Patients Over 55 Years of Age With Coronary Heart Disease in 6-min Walking Test in Cardiorespiratory Physiotherapy
Brief Title: Exploration of Possible Reasons for the Discrepancy Between Expectation and Indication of Subjective Perceived Exertions
Acronym: Ex-6-rate
Status: Completed | Type: Observational
Sponsor: Klinik Barmelweid (Other)
Responsible Party: Principal Investigator, Gilbert Busching, Physical Therapist, Klinik Barmelweid
Other Study IDs: 001
Record Dates: First submitted 2021-05-05; First posted 2021-05-24 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Coronary Disease; Exercise Test; Physical Exertion; Cardiac Rehabilitation; Physical Therapy
MeSH Terms: conditions — Coronary Disease | interventions — Surveys and Questionnaires; Interviews as Topic; Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients over 55 Years with coronary heart disease: Questionnaire and semistructured Interview 45 -60 minutes
  Interventions: Other: Questionnaire, Interview
- physical therapists working with patients with coronary heart disease: Focus group 60 -90 minutes
  Interventions: Other: Focus Group

INTERVENTIONS:
Other: Questionnaire, Interview — During the stay, a study visit is arranged with the patient after the 6-minute walk test has been performed. This consists of filling out the questionnaire and an interview, which lasts about 45-60 minutes. This is carried out by the investigator on at least 5 subjects. After each interview, a list of influencing factors is kept. If new aspects continue to appear in the 5th interview, the interviews are continued (up to a maximum of the 10th subject). If no new aspects appear in the interviews from number 6 onwards, the interviews are discontinued and no further patients are recruited. The conversations are recorded with an audio recording.
  Groups: Patients over 55 Years with coronary heart disease
Other: Focus Group — The focus group is carried out first in order to identify influencing variables that may be relevant for the interview (duration 60-90 minutes).
  Groups: physical therapists working with patients with coronary heart disease

SUMMARY:
The 6-minute walk test is a test of physical performance in physiotherapy with lungs and heart patients (Pollentier 2010). However, only 8 and 11% of patients in everyday test situations report a score of 7 or higher on a scale of 0-10 for effort (Jehn 2009). This study is intended to explore, based on grounded theory, why the majority of patients do not assess themselves according to the almost maximum performance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease undergoing in-patient cardiovascular rehabilitation; over 55 years of age. Patients underwent a 6-minute walk test with assessment of the intensity of the exercise

Exclusion Criteria:

* no understanding of the German language
* Patients would not be able to perform a 6-minute walk test, e. g. surgery on the large joints of the lower extremities, unstable heart disease or predominant neurological symptoms.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from the department of cardiology in the rehabilitation centre of Klinik Barmelweid AG,
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2022-08-14 (Actual)

PRIMARY OUTCOMES:
semi-structured interview about reasons, that could influence the rating of patients | during inpatient rehabilitation after the 1st six-minute-walking test within 3 weeks
  Patients were asked in a semi-structured interview about other reasons, that could influence their rating.
reasons, what might patients influence for ratings of patients given from physical therapist | with the beginning of the study within 4 weeks, before the patients' questionnaire and interview
  physical therapists identify reasons in a focus group, that influence the patients.

OTHER OUTCOMES:
Patients' experience with the conduction of the six-minute-walking test | during inpatient rehabilitation after the 1st six-minute-walking test within 3 weeks
  nominal scale (yes-partly-no)
Patients' honesty of the statement of effort | during inpatient rehabilitation after the 1st six-minute-walking test within 3 weeks
  nominal scale (yes-no)
Patients' exertion and performance limit | during inpatient rehabilitation after the 1st six-minute-walking test within 3 weeks
  open questions
Patients' safety during the six-minute-walking test | during inpatient rehabilitation after the 1st six-minute-walking test within 3 weeks
  numeric rating scale 0-10 (more likely no = 0; more likely yes = 10)
Patients' performance limit before and after the heart disease | during inpatient rehabilitation after the 1st six-minute-walking test within 3 weeks
  numeric rating scale 0-10 (more likely no = 0; more likely yes = 10)
Patients' sportiness | during inpatient rehabilitation after the 1st six-minute-walking test within 3 weeks
  numeric rating scale 0-10 (more likely no = 0; more likely yes = 10)
Experience of maximal exertion of activity in the past | during inpatient rehabilitation after the 1st six-minute-walking test within 3 weeks
  4-point nominal scale (weekly to several years ago)

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Büsching, Principal Investigator — Klinik Barmelweid AG
Locations (1):
- Klinik Barmelweid AG, Barmelweid, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jehn M, Halle M, Schuster T, Hanssen H, Weis M, Koehler F, Schmidt-Trucksass A. The 6-min walk test in heart failure: is it a max or sub-maximum exercise test? Eur J Appl Physiol. 2009 Oct;107(3):317-23. doi: 10.1007/s00421-009-1128-0. Epub 2009 Jul 18. PMID 19618202
- [Background] Pollentier B, Irons SL, Benedetto CM, Dibenedetto AM, Loton D, Seyler RD, Tych M, Newton RA. Examination of the six minute walk test to determine functional capacity in people with chronic heart failure: a systematic review. Cardiopulm Phys Ther J. 2010 Mar;21(1):13-21. PMID 20467515
- See also: Nationaler Verein für Qualitätsentwicklung in Spitälern und Kliniken. ANQ; Nationaler Vergleichsbericht 2018 - Kardiale Rehabilitation [Internet]. Messergebnisse Rehabilitation. 2018 [zitiert 7. Dezember 2020]. — http://results.anq.ch/fileadmin/documents/anq/27_31/20200424_ANQreha_Nationaler-Vergleichsbericht_2018_Kardiale-Rehabilitation.pdf